CLINICAL TRIAL: NCT01259063
Title: Phase I/II Study of RAD001 and Intravesical Gemcitabine in BCG-Refractory Primary or Secondary Carcinoma In Situ of the Bladder
Brief Title: RAD001 and Intravesical Gemcitabine in BCG-Refractory Primary or Secondary Carcinoma In Situ of the Bladder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry); New York University (Other); University of Hawaii (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-165
Record Dates: First submitted 2010-12-09; First posted 2010-12-13 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2017-06

CONDITIONS: Bladder Cancer
Keywords: GEMCITABINE; RAD001(EVEROLIMUS); urinary; BCG-Refractory; Intravesical; 10-165
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pts who failed or relapsed after intravesical BCG (Experimental): Phase I: Everolimus will be administered as follows: Dose level 1: 5 mg every other day, Dose level 2: 5 mg daily, Dose level 3: 10 mg daily Phase II: Everolimus will be administered at the dose determined in Phase .Everolimus will be continued for 12 months in the patients who achieve a CR or a Partial Response. Patients demonstrating a CR (by cystoscopy and cytology) or a Partial Response at their Cycle 12 cystoscopy will be observed with serial cystoscopies every 3 months.
  Interventions: Drug: Everolimus and Intravesical Gemcitabine

INTERVENTIONS:
Drug: Everolimus and Intravesical Gemcitabine — Phase I: Everolimus will be adm as follows: Dose level 1: 5 mg every other day, Dose level 2: 5 mg daily, Dose level 3: 10 mg daily Phase II: Everolimus will be adm at 10 mg daily the dose determined in Phase I. Pts will receive a dose of 2000 mg of intravesical gemcitabine twice a week (72-96 +8 hours between doses) for 3 weeks for a total of 6 treatments in course 1. After 1 week of rest from intravesical gemcitabine, course 2 will be administered, provided the treating physician notes acceptable pt tolerance. The total number of intravesical instillations will be 12. There will be no dose modifications to gemcitabine; however, pts will be allowed to skip gemcitabine doses if needed, per the treating physician's discretion. Missed or skipped doses of gemcitabine will not be repeated. The pt will receive as many instillations as tolerable up to the maximum of 12 instillations.

SUMMARY:
The purpose of this study is to test the safety of gemcitabine applied to the bladder directly combined with different oral doses of everolimus and to assess the right doses. Gemcitabine will be given at a fixed dose. Up to 3 dose levels of everolimus will be evaluated. The purpose of the phase II part is to test the combination of gemcitabine applied to the bladder directly combined with different oral doses of everolimus and to study the effects of these two drugs together. The investigators want to find out what effects, good and/or bad, this treatment has on the patient and the cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have Bacille Calmette-Guérin (BCG) refractory primary or secondary TisN0M0 BCG-refractory disease is defined as:
* Patient positive for Cis after 2 consecutive BCG installations
* OR, patient had a BCG response and failure within 6 months
* OR, patient has Cis on maintenance BCG
* OR, patient has persistent Cis 6 months after at least one instillation of BCG
* OR, patient is BCG intolerant
* OR, any of the above criteria for patients with a history of T1 disease
* OR, patient has BCG-relapsing disease, defined as failure more than 6 months after the patient was disease-free
* Pathologic confirmation of urothelial carcinoma by the enrolling institution
* Karnofsky Performance Status (KPS) ≥ 70%
* Age ≥ 18 years
* Adequate bone marrow function as shown by: ANC ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L, Hb >9 g/dL
* Adequate liver function as shown by:
* serum bilirubin ≤ 1.5 x ULN (upper limit of normal)
* ALT and AST ≤ 2.5x ULN
* International normalized ratio (INR) ≤1.5 x ULN (Anticoagulation is allowed if target INR ≤ 1.5 x ULN on a stable dose of warfarin or on a stable dose of low molecular weight (LMW) heparin for >2 weeks
* Adequate renal function: serum creatinine ≤ 1.5 x ULN
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid-lowering medication. After lipid-lowering therapy, patients must meet the same criteria, i.e. a fasting serum cholesterol < 300 mg/dL OR < 7.75 mmol/L AND fasting triglycerides < 2.5 x ULN, to be eligible for study treatment.
* Pre-treatment tumor tissue (minimum 10 slides) or 1 paraffin-embedded block when available for analysis of m-TOR pathway markers.
* Testing for hepatitis B viral load and serological markers (Hepatitis B PCR quantitative, HBsAg, HBsAb, and HBcAb) for the following patients:
* All patients who currently live in (or have lived in) Asia, Africa, Central and South America, Eastern Europe, Spain, Portugal, or Greece
* Patients with any of the following risk factors:
* Known or suspected past hepatitis B infection
* Blood transfusion(s) prior to 1990
* Current or prior IV drug users
* Current or prior dialysis
* Household contact with hepatitis B infected person(s)
* Current or prior high-risk sexual activity
* Body piercing or tattoos
* Mother known to have hepatitis B
* History suggestive of hepatitis B infection, e.g. dark urine, jaundice, or right upper quadrant pain
* Additional patients at the discretion of the site Principal Investigator
* Testing for hepatitis C infection (using quantitative RNA-PCR) for patients with any of the following risk factors:
* Known or suspected past hepatitis C infection (including patients with past interferon "curative" treatment)
* Blood transfusion(s) prior to 1990
* Current or prior IV drug users
* Household contact of hepatitis C infected person(s)
* Current or prior high-risk sexual activity
* Body piercing or tattoos
* Additional patients at the discretion of the site Principal Investigator

Exclusion Criteria:

* Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of study drug (including chemotherapy, radiation therapy, antibody based therapy, etc.) with the exception of topical anti-neoplastic agents that are not being used to treat malignancy
* Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery or patients that may require major surgery during the course of the study.
* Prior treatment with any investigational drug within the preceding 4 weeks
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
* Patients should not receive immunization with attenuated live vaccines within 1 week of study entry or during study period
* Other malignancies within the past 3 years, except for adequately treated carcinoma of the cervix, basal or squamous cell carcinomas of the skin or adenocarcinoma of the prostate that has been treated.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:
* symptomatic congestive heart failure of New York Heart Association Class III or IV
* unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease
* Severely impaired lung function as defined by spirometry and diffusing capacity of lung for carbon monoxide (DLCO) that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air
* uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN
* active (acute or chronic) or uncontrolled severe infections including urinary tract infections
* liver disease such as cirrhosis, chronic active hepatitis, or chronic persistent hepatitis
* A known history of HIV seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of Everolimus (eg, ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small-bowel resection)
* Patients with an active, bleeding diathesis
* Female patients who are pregnant or breast feeding, Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days prior to administration of Everolimus.
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing of study treatment. High effective contraception methods include combination of any two of the following (a+b or a+c or b+c):
* Use of oral, injected or implanted hormonal methods of contraception or;
* Placement of an intrauterine device (IUD) or intrauterine system (IUS);
* Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository;
* Total abstinence or;
* Male/female sterilization. Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to registration. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
* Male patients whose sexual partner(s) are WOCBP who are not willing to use adequate contraception during the study and for 8 weeks after the end of treatment.
* Patients with a known hypersensitivity to Everolimus or other rapamycins (sirolimus, temsirolimus) or to its excipients
* History of noncompliance to medical regimens
* Patients unwilling to or unable to comply with the protocol
* Prior radiation to the pelvis for bladder cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guido Dalbagni, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Everolimus and Intravesical Gemcitabine: Phase I: Everolimus will be administered as follows: Dose level 1: 5 mg every other day, Dose level 2: 5 mg daily, Dose level 3: 10 mg daily Phase II: Everolimus will be administered at the dose determined in Phase .Everolimus will be continued for 12 months in the patients who achieve a CR or a Partial Response.
Period: Overall Study
Arm/Group | Everolimus and Intravesical Gemcitabine
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pts Who Failed or Relapsed After Intravesical BCG
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: years] | 66 [49 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Phase I - Dose-limiting Toxicity (DLT)
Description: Everolimus (mg) given in conjunction with intravesical gemcitabine
Time Frame: 8 weeks
Population: 14 of the 33 participants were enrolled in the Phase I portion of the protocol
Measure: Number; unit: DLT
Groups:
- Pts Who Failed or Relapsed After Intravesical BCG: Phase I: Everolimus will be administered as follows: Dose level 1: 5 mg every other day, Dose level 2: 5 mg daily, Dose level 3: 10 mg daily Phase II: Everolimus will be administered at the dose determined in Phase I.
Arm/Group | Pts Who Failed or Relapsed After Intravesical BCG
Number analyzed (Participants) | 14
DLT | 0

2. Primary Outcome: Phase II - Patients Who Are Free of Disease at 1 Year
Description: following start of therapy.
Time Frame: 1 year
Population: 19 participants were evaluable for Phase II.
Measure: Number (95% Confidence Interval); unit: percentage of pts disease free at 1 year
Arm/Group | Pts Who Failed or Relapsed After Intravesical BCG
Number analyzed (Participants) | 19
percentage of pts disease free at 1 year | 21 [0 to 43]

3. Primary Outcome: Phase I - Maximum Tolerated Dose (MTD)
Description: of Everolimus given in conjunction with intravesical gemcitabine
Time Frame: 8 weeks
Population: 14 participants enrolled in Phase I
Measure: Number; unit: mg daily of everolimus
Arm/Group | Pts Who Failed or Relapsed After Intravesical BCG
Number analyzed (Participants) | 14
mg daily of everolimus | 10

4. Secondary Outcome: Complete Response (CR) Rate
Description: Complete Response (CR) is defined as no evidence of disease (by cytology and cystoscopy). Partial Response is defined as negative cystoscopy and positive cytology. Progression is defined as the development of invasion or metastasis. If the participant develops a recurrence, they will be considered having failed treatment. Participants will also be considered having failed treatment if there is no response to treatment after two cycles.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pts Who Failed or Relapsed After Intravesical BCG
Number analyzed (Participants) | 33
Participants
  Complete Response | 17
  Partial Response | 8
  Did not achieve CR or PR | 8

5. Secondary Outcome: Survival of Patients Treated
Description: With Everolimus in combination with intravesical gemcitabine. Overall survival following start of therapy will be estimated using Kaplan-Meier methods.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: % of pts with CR who relapsed in a year
Arm/Group | Pts Who Failed or Relapsed After Intravesical BCG
Number analyzed (Participants) | 33
% of pts with CR who relapsed in a year | 21 [0 to 43]

6. Secondary Outcome: Activated mTOR (Mammalian Target of Rapamycin) Pathway Markers as Well as Phosphatase and Tensin Homolog (PTEN) Status and Serine/Threonine Kinase (AKT) Activation Evaluation
Description: In all pre-treatment specimens and analysis of post treatment specimens when available.
Time Frame: 1 year
Population: Inability for sequencing due to inadequate amount of tissue
Arm/Group | Pts Who Failed or Relapsed After Intravesical BCG
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Pts Who Failed or Relapsed After Intravesical BCG
All-Cause Mortality (participants affected / at risk) | 4/33
Serious Adverse Events (participants affected / at risk) | 13/33
Other Adverse Events (participants affected / at risk) | 23/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pts Who Failed or Relapsed After Intravesical BCG (N=33)
Abdominal distension (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Anemia (Blood and lymphatic system disorders) | 2
Aspartate aminotransferase increased (Investigations) | 1
Chills (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Ejection fraction decreased (Investigations) | 1
Fever (General disorders) | 3
Gastric ulcer (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Gen disorders & admin site conditions Other, spec (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Injury/poison & proced complications Other, spec (Injury, poisoning and procedural complications) | 1
Myocardial infarction (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pts Who Failed or Relapsed After Intravesical BCG (N=33)
Hyperglycemia (Metabolism and nutrition disorders) | 22
Alanine aminotransferase increased (Investigations) | 19
Cholesterol high (Investigations) | 18
Aspartate aminotransferase increased (Investigations) | 17
Hypertriglyceridemia (Metabolism and nutrition disorders) | 17
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 16
Anemia (Blood and lymphatic system disorders) | 14
Fatigue (General disorders) | 12
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 12
Mucositis oral (Gastrointestinal disorders) | 11
Platelet count decreased (Investigations) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Hypernatremia (Metabolism and nutrition disorders) | 9
Diarrhea (Gastrointestinal disorders) | 8
Dysgeusia (Nervous system disorders) | 8
Headache (Nervous system disorders) | 8
Hypoalbuminemia (Metabolism and nutrition disorders) | 8
White blood cell decreased (Investigations) | 8
Alkaline phosphatase increased (Investigations) | 7
Creatinine increased (Investigations) | 7
Dry skin (Skin and subcutaneous tissue disorders) | 6
Hyperkalemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 6
Urinary frequency (Renal and urinary disorders) | 6
Edema limbs (General disorders) | 5
Endocrine disorders - Other, specify (Endocrine disorders) | 5
Erythema multiforme (Skin and subcutaneous tissue disorders) | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Skin & subcutaneous tissue disorders Other, spec (Skin and subcutaneous tissue disorders) | 5
Weight loss (Investigations) | 5
Burn (Injury, poisoning and procedural complications) | 4
Cystitis noninfective (Renal and urinary disorders) | 4
Fever (General disorders) | 4
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 4
Blood bilirubin increased (Investigations) | 3
Dry mouth (Gastrointestinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Hematuria (Renal and urinary disorders) | 3
Lymphocyte count decreased (Investigations) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Flu like symptoms (General disorders) | 2
Gen disorders & admin site conditions Other, spec (General disorders) | 2
Hypertension (Vascular disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
INR increased (Investigations) | 2
Nausea (Gastrointestinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 2
Urinary tract pain (Renal and urinary disorders) | 2
Urinary urgency (Renal and urinary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2011-01-11): https://cdn.clinicaltrials.gov/large-docs/63/NCT01259063/Prot_000.pdf
  • Informed Consent Form (2011-01-11): https://cdn.clinicaltrials.gov/large-docs/63/NCT01259063/ICF_001.pdf
  • Statistical Analysis Plan (2018-01-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT01259063/SAP_002.pdf